CLINICAL TRIAL: NCT05379010
Title: Endodontic Microsurgery With the Use of L-PRF Block: a Randomized Controlled Clinical Trial
Brief Title: Endodontic Microsurgery With the Use of L-PRF Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S63971
Record Dates: First submitted 2022-04-22; First posted 2022-05-18 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Apical Periodontitis; Apical Periodontal Cyst
MeSH Terms: conditions — Periapical Periodontitis; Radicular Cyst

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With L-PRF Block (Experimental)
  Interventions: Procedure: Endodontic Microsurgery
- No L-PRF Block (Active Comparator)
  Interventions: Procedure: Endodontic Microsurgery

INTERVENTIONS:
Procedure: Endodontic Microsurgery — Surgical removal of 3 millimeters of the root-end, removal of the apical pathology, Root-end preparation and retrograde filling. The entire procedure is done under magnification.

SUMMARY:
This study evaluates the effect of leucocyte and platelet rich fibrin Block (L-PRF Block) during endodontic microsurgery (EMS) on patient's post-operative comfort and periapical bone healing in large peri-apical lesions.

DETAILED DESCRIPTION:
This study evaluates the effect of leucocyte and platelet rich fibrin Block (L-PRF Block) during endodontic microsurgery (EMS) on patient's post-operative comfort and periapical bone healing in large peri-apical lesions. The trial design is an open randomized controlled clinical trial with two groups. Half of the participants will receive EMS with L-PRF Block (experimental group), the other half without (control group).

ELIGIBILITY:
Inclusion Criteria

* Provision of Informed Consent
* Patients from 18 years old
* Patients in need of an EMS
* EMS is the only option to cure the periapical lesion
* A periapical lesion that has a diameter of 10mm or more in sagittal plane, frontal plane or axial plane when measured on CBCT

Exclusion Criteria

* Unlikely to be able to comply with the study procedures, as judged by the investigator
* Orthograde endodontic (re)treatment is indicated
* Known or suspected current malignancy
* History of chemotherapy within 5 years prior to study
* History of radiation in the head and neck region
* History of other metabolic bone diseases
* History of bleeding disorders
* HIV disease
* Hepatitis B or C
* Systemic disease (osteoporosis, diabetes…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Amount of peri-apical bone healing | 1 year
  Amount of periapical bone healing in time: measured with Cone Beam Computed Tomography (CBCT).

SECONDARY OUTCOMES:
Patient related outcomes | 7 days
  Pain assessed with a Visual Analogue Scale ranging from 0 to 10 each day during the first 7 days post-op.
Patient related outcomes | 7 days
  Pain assessed with a questionnaire asking about analgesics usage each day during 7 days post-op.
Patient related outcomes | 7 days
  Discomfort assessed with a Visual Analogue Scale ranging from 1 to 5 each day during the first 7 days post-op.
Bone or scar tissue healing | 1 year
  Bone or scar tissue healing: Volumetric analysis using Cone-Beam Computed Tomography. Pre-operative CBCT data will be matched with the post-op CBCT scans in order to assess the volumetric changes during 1 year.
Success & survival rate | 1 year
  Success & survival rate
Dentinal defects | 1 year
  Dentinal defects: in the apical root before and after resection. Potential cracks and fractures that occur during the follow-up period will be assessed on CBCT en reported.

CONTACTS AND LOCATIONS:
Overall Officials: Nastaran Meschi, DDS, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No